CLINICAL TRIAL: NCT00717743
Title: T Regulatory Cells in Renal Cell Carcinoma (PILOT STUDY)
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: RC02/31/06
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2010-04

CONDITIONS: Renal Cell Carcinoma
Keywords: RCC; patients; scheduled; nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Patients diagnosed with RCC.

SUMMARY:
To define the frequency of T regulatory cells in peripheral blood of RCC patients before and after nephrectomy.

Study hypothesis: That nephrectomy results in a normalisation of peripheral blood T regs in early stage RCC, and a lowering of T regs in advanced RCC.

DETAILED DESCRIPTION:
T regulatory cells (T regs) are a recently identified subset of T cells with inhibitory functions on the immune system. In cancer, it has been shown that there is an increased proportion of T regs in several different human malignancy states. T regs are found to be elevated in peripheral blood mononuclear cells, draining lymph nodes and in the primary tumor itself. There has also been correlation between peripheral blood T regs and tumor stage, tumor relapse and survival. It has been proposed that the T regs are activated and expanded by factors produced by the tumor microenvironment. They are thought to play a role in preventing or demising host T-cell responses against cancer, including a suboptimal host responses to vaccine strategies. Strategies to reduce T regs in cancer patients are being explored as a novel immunologic anti-cancer approach.

Renal cell cancer (RCC) is a tumor with well-known immune-mediated phenomena such as spontaneous regression. There is paucity of data on T regs in RCC. We propose to study the frequency of peripheral blood T regs before and after nephrectomy for RCC. We will document the baseline frequency of T regs in RCC and if nephrectomy results in a change in levels. We hypothesize that nephrectomy will lower peripheral T regs to normal levels in early stage RCC, and will reduce peripheral T reg levels in advanced RCC patients. If found to be so, T regs could in future be used as an indicator of disease recurrence in early stage RCC. In advanced RCC, lowering of T reg levels may help explain the previous hypothesis that debulking nephrectomy results in improved anti-tumor immunity, provide rationale for second debulking procedures, and be correlated with subsequent clinical course.

The main laboratory technique is flow cytometry. This will be a pilot study with small patient numbers. Only blood samples are required.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the inclusion criteria to participate in this study:

* Diagnosed Renal Cell Carcinoma patients for whom nephrectomy is planned or scheduled as treatment. (Preoperative histologic diagnosis is not required.)
* All stages of disease are eligible.
* Adult patients above 21.
* Ability to provide informed consent

Exclusion Criteria:

Subjects meeting any of the exclusion criteria at baseline will be excluded:

* Active infection.
* Immunocompromised or other active immune disorders.
* Not on any immunomodulating therapy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RCC patients scheduled for nephrectomy
Sampling Method: Probability Sample
Dates: Start 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: Alvin Seng Cheong Wong, MBBS, MRCP, Principal Investigator — National University Hospital, Singapore; Chin Tiong Heng, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- National University Hospital, Singapore, Singapore